CLINICAL TRIAL: NCT05464537
Title: To Assess the Efficacy Rate of Unipolar Polarity Switch for Lesion Assessment in Pulmonary Vein Isolation
Brief Title: Efficacy Rate of Unipolar Polarity Switch for Lesion Assessment in Pulmonary Vein Isolation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company which provides funding is closed
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Collaborators: Kansas City Heart Rhythm Institute, Overland Park, KS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KCHRRF-UNIPOLAR SWITCH-0013
Record Dates: First submitted 2022-07-06; First posted 2022-07-19 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unipolar Polarity Switch Left and CAI-OPR-LAAP Right (Active Comparator)
  Interventions: Other: Unipolar Polarity Switch Left
- CAI-OPR-LAAP Left and Unipolar Polarity Switch Right (Active Comparator)
  Interventions: Other: Unipolar Polarity Switch Right

INTERVENTIONS:
Other: Unipolar Polarity Switch Left — 10-15 Left veins are randomized to Unipolar Polarity Shift, right veins are randomized to CAI-OPR-LAAP
  Arms: Unipolar Polarity Switch Left and CAI-OPR-LAAP Right
Other: Unipolar Polarity Switch Right — 10-15 cases randomized to CAI-OPR-LAAP on left veins, and Unipolar Polarity Switch on right veins
  Arms: CAI-OPR-LAAP Left and Unipolar Polarity Switch Right

SUMMARY:
The technique of intraprocedural electrogram morphology as a measure of lesion effectiveness in an attempt to achieve durable PVI, clearly led to shortened procedural time, radiation exposure, and superiority in outcomes, with the implementation of a reproducible, readily available intraprocedural tool that can be applied universally.

DETAILED DESCRIPTION:
One initial study reported that unipolar atrial EGM modification was a useful end point for RF energy delivery. They compared 2 groups of patients with paroxysmal AF undergoing PVI facilitated by an electroanatomic mapping system, merged preprocedural LA computed tomographic scan, and a circular mapping catheter.

They were the first to use intraprocedural electrogram morphology as a measure of lesion effectiveness in an attempt to achieve durable PVI. The technique, clearly led to shortened procedural time, radiation exposure, and superiority in outcomes, with the implementation of a reproducible, readily available intraprocedural tool that can be applied universally.

As there is scant data is this area with lack of randomized human trials, planned on building and further validating evidence from Bortone et al in demonstrating that loss of unipolar negative component during PVI can serve a great adjuvant tool for achieving durability of PVI with overall lesser procedural time and no significant increase in adverse events.

ELIGIBILITY:
Inclusion Criteria:

* All Patients ≥ 18 years of age
* Undergoing pulmonary vein isolation for De-Novo Atrial Fibrillation.

Exclusion Criteria:

* Patients unable to give consent
* Who do not have De-novo AF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Efficacy rate of loss of unipolar negative component | Procedure day and 12 month follow-up day
  Observe the efficacy rate of loss of unipolar negative component in isolation of the Pulmonary Veins. Loss of unipolar negative component will be assessed during the Radiofrequency ablation procedure. The durability of Pulmonary vein isolation will be assessed at 12 month follow up, if there is recurrence of Atrial fibrillation.
Number of patients with Esophageal Injury | 1 year
  Number of patients with intraprocedural and post procedure adverse events and serious adverse events - Esophageal Injury
Number of patients with TIA/CVA | 1 year
  Number of patients with intraprocedural and post procedure adverse events and serious adverse events - transient ischemic attack/Cerebrovascular accident (TIA/CVA)
Number of patients with Bleeding/Hematoma | 1 year
  Number of patients with intraprocedural and post procedure adverse events and serious adverse events - Bleeding/Hematoma
Number of patients with Pericardial Effusion | 1 year
  Number of patients with intraprocedural and post procedure adverse events and serious adverse events - Pericardial Effusion
Number of patients with need for open heart surgery | 1 year
  Number of patients with intraprocedural and post procedure adverse events and serious adverse events - need for open heart surgery
Number of patients with phrenic nerve injury | 1 year
  Number of patients with intraprocedural and post procedure adverse events and serious adverse events - phrenic nerve injury
Number of patients with pulmonary vein stenosis | 1 year
  Number of patients with intraprocedural and post procedure adverse events and serious adverse events - pulmonary vein stenosis
Esophageal Temp max (existing protocol) | 1 day
  Esophageal temp max (existing protocol)
Esophageal "Time above threshold" | 1 day
  Esophageal "Time above threshold"
Esophageal "Time to return to baseline" | 1 day
  Esophageal "Time to return to baseline"
Images comparing PURE EP unipolar signals against Claris unipolar signals | 1 day
  Observe if the quality of PURE EP's unipolar signals are acutely and better suited for lesion assessment? This outcome compares mapping images with site of activation to the PURE EP electrogram and compare if they correspond to each other.

SECONDARY OUTCOMES:
Compare 1st pass isolation | 1 day
  Compare 1st pass isolation in the Unipolar polarity switch group to Carto's Ablation Index per Overland Park Regional's Left Atrial Ablation Protocol (CAI-OPR-LAAP)
Total RF Time | 1 day
  Total RF Time in pulmonary veins with Unipolar polarity switch as endpoint vs. CAI-OPR-LAAP
Discrimination with High Frequency Algorithm as a confirmation tool | 1 day
  In Left Superior Vein, Right Superior Vein, and Right Inferior Vein, validate Near Field and Far Field Discrimination with High Frequency Algorithm as a confirmation tool (Visitag #'s annotated into PURE EP)
6-month freedom from AF | 6 months
  6-month freedom from AF
Redo's within 1 year | 1 year
  Redo's within 1 year which vein randomized group reconnected
Location of Catheter tip | 1 day
  Location of Catheter tip (LSPV, RSPV, RIPV, LIPV, LAA, Other) (carto image)
Duration of HFA channel compared to Bipolar | 1 day
  Duration of HFA channel compared to Bipolar, Was there both a near and far field component?

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (2):
- United States (2):
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bortone A, Brault-Noble G, Appetiti A, Marijon E. Elimination of the negative component of the unipolar atrial electrogram as an in vivo marker of transmural lesion creation: acute study in canines. Circ Arrhythm Electrophysiol. 2015 Aug;8(4):905-11. doi: 10.1161/CIRCEP.115.002894. Epub 2015 Jun 19. PMID 26092576
- [Background] Pambrun T, Durand C, Constantin M, Masse A, Marra C, Meillet V, Haissaguerre M, Jais P, Bortone A. High-Power (40-50 W) Radiofrequency Ablation Guided by Unipolar Signal Modification for Pulmonary Vein Isolation: Experimental Findings and Clinical Results. Circ Arrhythm Electrophysiol. 2019 Jun;12(6):e007304. doi: 10.1161/CIRCEP.119.007304. Epub 2019 Jun 5. PMID 31164003
- [Background] Bortone A, Appetiti A, Bouzeman A, Maupas E, Ciobotaru V, Boulenc JM, Pujadas-Berthault P, Rioux P. Unipolar signal modification as a guide for lesion creation during radiofrequency application in the left atrium: prospective study in humans in the setting of paroxysmal atrial fibrillation catheter ablation. Circ Arrhythm Electrophysiol. 2013 Dec;6(6):1095-102. doi: 10.1161/CIRCEP.113.000749. Epub 2013 Oct 4. PMID 24097371